A single center randomized prospective study on the peristaltic direction of gastrointestinal anastomosis in Roux-en-Y reconstruction after distal curative gastrectomy for gastric cancer (DJY002 Trail)

**Edition Number: 1.0** 

**Edition Generation Date: Qct 30, 2020** 

Principal Investigator: Jingyu Deng and Han Liang

Research Institute: Cancer Hospital & Institute of Tianjin Medical University

## **Statistical Analysis Plan**

Continuous variables are presented as mean  $\pm$  standard deviation or median (interquartile range). Statistical analyses were performed using the chi-square test for the categorical variables and the Mann–Whitney U-test for the continuous variables. Multivariable analysis to identify relationships among clinicopathological variables was carried out by means of multinomial logistic regression. The time of early recovery postoperatively in relation to different peristaltic direction of gastrointestinal anastomosis was evaluated by Kaplan–Meier analysis and log rank test. Cox proportional hazards model was used for multivariable analysis. A p-value threshold of 0.05 was considered statistically significant. All statistical analyses were performed using PASW 18.0 software.